CLINICAL TRIAL: NCT01908855
Title: Enriching Cognitive-Behavioral Therapy With Emotion Regulation Training in Patients With Chronic Multiple Somatoform Symptoms (ENCERT): A Randomized Controlled Trial
Brief Title: Cognitive-Behavioral Therapy Enriched With Emotion Regulation Training for Multiple Somatoform Symptoms
Acronym: ENCERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: University of Technology Munich (Unknown); Central Institute of Mental Health, Mannheim (Other); University of Giessen (Other); University of Wuppertal (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University of Kaiserslautern-Landau (Other); German Research Foundation (Other); Philipps University Marburg Coordination Centre for Clinical Trials (Unknown)
Responsible Party: Principal Investigator, Winfried Rief, Professor of Clinical Psychology, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENCERT-130313; Ri 574/24-1 (Other Grant/Funding Number: German Research Foundation DFG)
Record Dates: First submitted 2013-07-19; First posted 2013-07-26 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Somatic Symptom Disorder (DSM-V)
Keywords: somatoform symptoms; somatic symptoms; somatoform disorder; somatic symptom disorder; cognitive-behavioral therapy; emotion regulation training
MeSH Terms: conditions — Medically Unexplained Symptoms; Somatoform Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENCERT (Experimental): ENCERT contains 1) psychoeducation (session1), 2) relaxation techniques for coping with stress (sessions 2-4), 3) non-judgmental awareness of body perceptions, (sessions 5-7), 4) modifying illness behavior and accepting unpleasant body perceptions (sessions 8-13), 5) attention defocusing on positive perceptions plus emotional self-support (sessions 14- 15), 6) analyzing interpretation processes to understand situational cues (sessions 16-17), and 7) change of behavior and interpretations (sessions 18-20). The innovative elements of ENCERT are: improving the awareness for the association of somatic symptoms with emotions, learning non-judgmental awareness and acceptance of unpleasant body perceptions, achieving high-frequent skill exercising with the emotion regulation audio training.
  Interventions: Behavioral: Cognitive-behavioral therapy + emotion regulation training for patients with multiple somatoform symptoms
- CBT (Active Comparator): This arm is based on traditional cognitive-behavioral therapy that can be considered the current "treatment of choice", being the only intervention with an evidence grade 1a (Kroenke, 2007). As such, it presents the reference of efficacy and safety for new regimen. The strictly manualized program includes the following components focusing on the special needs of chronic somatoform patients: psychoeducation providing a framework for psychotherapy, attention defocusing, reduction of over-interpretation of symptoms, increase of physical activity, stress reduction.
  Interventions: Behavioral: Cognitive-behavioral therapy for patients with multiple somatoform symptoms

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy + emotion regulation training for patients with multiple somatoform symptoms — Cognitive-behavioral therapy + emotion regulation training for patients with multiple somatoform symptoms:
  20 weekly sessions individual therapy (à 50) minutes
  Arms: ENCERT
Behavioral: Cognitive-behavioral therapy for patients with multiple somatoform symptoms — Cognitive-behavioral therapy for patients with multiple somatoform symptoms:
  20 weekly sessions individual therapy (à 50) minutes
  Arms: CBT

SUMMARY:
The purpose of this study is to evaluate whether cognitive-behavioral therapy enriched with strategies from emotion regulation training leads to better improvement in somatic symptoms and comorbid problems than cognitive-behavioral therapy alone.

DETAILED DESCRIPTION:
Somatic symptoms not caused by a known biomedical condition ("somatoform disorders") are highly prevalent, involve a high risk of chronicity, are one of the major reasons for doctor visits, and are a tremendous burden for health care systems. Despite the economic relevance, research activities are disproportionately low. The only intervention with an evidence grade I is cognitive-behavioral therapy (CBT). However, average effect sizes for CBT in somatization syndromes are only moderate (Cohen's d < 0.5), and more powerful interventions are needed.

There is convincing evidence that patients with somatoform disorders have emotion regulation deficits, which are not addressed by current CBT approaches. Based on positive results of a small pilot study it is expected that enriching CBT programs with emotion regulation techniques improves treatment outcome. The primary goal of the proposed project is therefore to evaluate this hypothesis in a randomized design.

Patients will be primarily recruited via referrals by primary care doctors. After a screening phase a baseline assessments with different self- and clinician-rating scales (see Outcome Measures) follows. If participants fulfill the eligibility criteria they will be randomized to one of the two study arms: cognitive-behavioral therapy vs. cognitive-behavioral therapy enriched with emotion regulation strategies. After every therapy session patients will be screened in regard to aspects of therapeutic alliance, adverse events, and symptom intensity/annoyance. The post assessment takes place after the 20th session and a follow-up is planned six months after post treatment.

Different methods will be applied to prevent bias and to assure a high quality level of the current study. Data handling, data monitoring and statistical analyses will be supervised by the Coordinating Center for Clinical Trials (KKS) of Philipps-University of Marburg; data quality and safety principles will be applied. Additionally an independent Data Safety Monitoring Board will be nominated. The study center will visit all study sites regularly to verify correct procedures, data sampling, and data management. Randomisation occurs and is controlled centrally through the randomisation's central office in KKS Marburg. Furthermore the current study constitutes a single-blinded trial. Assessment interviews are conducted and analyzed by people blinded to the treatment condition. Additionally, treatments are manualized, and therapists receive an intense training. Treatment fidelity/integrity is analyzed with rating schemes for 5% randomly selected videotaped treatment sessions. Allowed additional treatments during study inclusion are thoroughly monitored and analyzed.

The sample size calculation is based on the primary outcome variable "somatization severity index" of the Screening of Somatoform Disorders (SOMS-7T). Based on results of the main validation study of SOMS-7T, meta-analytic estimations, and results of a pilot study of the efficacy of ENCERT, the power calculations yield a necessary total sample size of N=194 to detect a clinical relevant difference of 4 points symptom reduction on SOMS-7T between the two treatments with a power of 0.80 and an alpha=.05. With regard to an estimated drop-out rate of 20%, N=244 patients are to be recruited.

As main efficacy analysis the primary outcome shall be analyzed with linear mixed-effect models. It will be done according to the Intention-to-Treat (ITT) principle: to consider missing values as a potential source of bias, they will be handled according to the framework by Rubin. Secondary statistical analyses focus on establishing longer term treatment efficacy and describing the pattern of change. For this purpose the mean response will be modeled as a function of time with a separate mixed effects linear model over all assessments. Furthermore, interindividual differences in intraindividual change will be modeled using multilevel analysis for longitudinal data. Multilevel longitudinal mediation analyses will be conducted in order to test whether the effect of treatment condition on intraindividual changes in somatic symptom severity can be explained by intraindividual changes in emotion regulation skills.

ELIGIBILITY:
Inclusion Criteria (are based on DSM-V diagnosis "somatic symptom disorder [SSD] 300.82"):

* Multiple distressing somatic symptoms (≥ 3 symptoms) not fully explained by a medical condition
* PDI ≥ 4
* Patient Health Questionnaire-15 (PHQ-15) ≥ 5
* Requested psychological criteria for SSD (at least 1 of 3):

  1. Disproportionate and persistent thoughts about the seriousness of one's symptoms
  2. Persistently high level of anxiety about health or symptoms
  3. Excessive time and energy devoted to these symptoms or health concerns
* Symptom duration ≥ 6 months
* Age: 18-69 years
* Comorbidity (depression, other mental disorders) allowed, as long as somatic symptoms are considered to be the major problem by therapist and patient
* Thorough medical check for medical disease that might fully explain the somatic symptoms
* Documented medical evaluation

Exclusion Criteria:

* Severe alcohol/drug addiction
* Acquired brain injuries
* Psychoses (history of schizophrenia spectrum disorders; bipolar disorders)
* Primary disorder requesting other treatments (e.g., suicidality)
* Biomedical etiology of major symptoms (also if detected during treatment course
* Ongoing psychotherapy
* Continuous or intermittent, high-dosage (on average more than once per 2 weeks) benzodiazepine treatment
* Continuous antipsychotic treatment
* Continuous opioid treatment
* For patients on medication with antidepressants: treatment regime changes during the time between 4 weeks prior to treatment until follow-up

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in somatic symptom severity (Screening of Somatoform Disorders, SOMS-7T) from pre-assessment to four in-between assessments to post-assessment to follow-up | From pre-assessment (admission) to four in-between assessments (9, 13, 17, 21 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of somatic symptom severity during the last 7 days (self-rating)

SECONDARY OUTCOMES:
Change in depressive symptoms (Beck Depression Inventory-II, BDI-II) from pre-assessment to one in-between assessment to post-assessment to follow-up | From pre-assessment (admission) to one in-between assessment (13 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of depressive symptoms (self-rating)
Change in emotion regulation skills (Emotion Regulation Skills Questionnaire, ERSQ) from pre-assessment to one in-between assessment to post-assessment to follow-up | From pre-assessment (admission) to one in-between assessment (13 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of emotion regulation skills (self-rating)
Change in symptom-focussed coping strategies (Pain Coping Questionnaire, FESV; Geissner, 2003) from pre-assessment to one in-between assessment to post-assessment to follow-up | From pre-assessment (admission) to one in-between assessment (13 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of symptom-focused coping strategies (self-rating)
Change in general psychopathological symptoms (Symptom Checklist-90, SCL-90) from pre-assessment to one in-between assessment to post-assessment to follow-up | From pre-assessment (admission) to one in-between assessment (13 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of general psychopathological symptoms (self-rating)
Change in symptom-caused disability (Pain Disability Index, PDI) from pre-assessment to one in-between assessment to post-assessment to follow-up | From pre-assessment (admission) to one in-between assessment (13 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of symptom-caused disability in different areas of life (self-rating)
Change in health-related quality of life (EuroQoL-5D, EQ-5D) from pre-assessment to one in-between assessment to post-assessment to follow-up | From pre-assessment (admission) to one in-between assessment (13 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of health-related quality of life (self-rating)
Change in health anxiety (Whiteley Index, WI) from pre-assessment to one in-between assessment to post-assessment to follow-up | From pre-assessment (admission) to one in-between assessment (13 weeks after admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Assessment of health anxiety (self-rating)
Change in social competence, emotion regulation, relaxation abilities, stress management, etc., in different areas of life (The Operationalized Assessment of Abilities, OFD) from pre-assessment to post-assessment to follow-up | From pre-assessment (admission) to post-assessment (25 weeks after admission) to follow-up (12 months after admission)
  Observer-based assessment of scores for social competence, emotion regulation, relaxation abilities, stress management, etc., in different areas of life (job, family, leisure)
Change in health care utilization and indirect costs (Structured Interview for the Assessment of Health Care Utilization, HCU) from pre-assessment to follow-up | From pre-assessment (admission) to follow-up (12 months after admission)
  Observer-based assessment of HCU and indirect costs. HCU will be transformed to costs using health economy tables
Inventory of the Assessment of Negative Effects of Psychotherapy (INEP) at post-assessment | Post-assessment (25 weeks after admission)
  Assessment of psychotherapy-induced side effects (self-rating)
Inventory of the Assessment of Negative Effects of Psychotherapy (INEP) at follow-up | Follow-up (12 months after admission)
  Assessment of psychotherapy-induced side effects (self-rating)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Ph.D., Principal Investigator — Philipps University Marburg; Mathias Berking, Ph.D., Study Chair — Philipps University Marburg; Maria Kleinstäuber, Ph.D., Study Chair — Philipps University Marburg; Japhia-Maria Gottschalk, M.Sc., Study Chair — Philipps University Marburg
Locations (7):
- Germany (7):
  - Justus-Liebig-University, CBT Outpatient Clinic, Giessen
  - University Medical Center Hamburg-Eppendorf, Department of Psychosomatic Medicine, Hamburg
  - University Koblenz-Landau, Department of Clinical Psychology and Psychotherapy, Koblenz-Landau
  - Central Institute of Mental Health, Department of Clinical Psychology, Mannheim
  - Philipps-University, Department of Clinical Psychology and Psychotherapy, Marburg
  - Rechts der Isar Hospital, University of Technology, Department of Psychosomatic Medicine and Psychotherapy, München
  - Bergische University, Department of Clinical Psychology and Psychotherapy, Wuppertal

REFERENCES:
- [Background] Barsky AJ, Orav EJ, Bates DW. Somatization increases medical utilization and costs independent of psychiatric and medical comorbidity. Arch Gen Psychiatry. 2005 Aug;62(8):903-10. doi: 10.1001/archpsyc.62.8.903. PMID 16061768
- [Background] Geissner E. Pain Coping Questionnaire FESV. Göttingen, Germany: Hogrefe; 2003.
- [Background] Göllner R, Gollwitzer M, Heider J, Zaby A, Schröder A. Analyzing longitudinal data with hierarchical linear models. Zeitschrift für Klinische Psychologie und Psychotherapie 39(3):179-88, 2010.
- [Background] Gottschalk JM, Bleichhardt G, Kleinstäuber M, Berking M, Rief W. Treatment efficacy of multiple somatoform symptoms? Enriching cognitive behavioral therapy with emotion regulation training: Results of a controlled pilot study. In preparation.
- [Background] Jacobi F, Wittchen H-U, Holting C, Hofler M, Pfister H, Muller N, Lieb R. Prevalence, co-morbidity and correlates of mental disorders in the general population: results from the German Health Interview and Examination Survey (GHS). Psychol Med. 2004 May;34(4):597-611. doi: 10.1017/S0033291703001399. PMID 15099415
- [Background] Kleinstauber M, Witthoft M, Hiller W. Efficacy of short-term psychotherapy for multiple medically unexplained physical symptoms: a meta-analysis. Clin Psychol Rev. 2011 Feb;31(1):146-60. doi: 10.1016/j.cpr.2010.09.001. Epub 2010 Sep 16. PMID 20920834
- [Background] Kroenke K. Efficacy of treatment for somatoform disorders: a review of randomized controlled trials. Psychosom Med. 2007 Dec;69(9):881-8. doi: 10.1097/PSY.0b013e31815b00c4. PMID 18040099
- [Background] Molenberghs G, Kenward MG.Missing Data in Clinical Studies. Chichester, UK: Whiley; 2007.
- [Background] Moscovitch DA, Hofmann SG, Suvak MK, In-Albon T. Mediation of changes in anxiety and depression during treatment of social phobia. J Consult Clin Psychol. 2005 Oct;73(5):945-952. doi: 10.1037/0022-006X.73.5.945. PMID 16287394
- [Background] Rief W, Hiller W. A new approach to the assessment of the treatment effects of somatoform disorders. Psychosomatics. 2003 Nov-Dec;44(6):492-8. doi: 10.1176/appi.psy.44.6.492. PMID 14597684
- [Background] Rief W, Rojas G. Stability of somatoform symptoms--implications for classification. Psychosom Med. 2007 Dec;69(9):864-9. doi: 10.1097/PSY.0b013e31815b006e. PMID 18040096
- [Background] Rieffe C, Terwogt MM, Bosch JD, Kneepkens CMF, Douwes AC, Jellesma FC. Interaction between emotions and somatic complaints in children who did or did not seek medical care. Cognition Emotion 21(8):1630-1646, 2007.
- [Background] Waller E, Scheidt CE. Somatoform disorders as disorders of affect regulation: a study comparing the TAS-20 with non-self-report measures of alexithymia. J Psychosom Res. 2004 Sep;57(3):239-47. doi: 10.1016/S0022-3999(03)00613-5. PMID 15507250
- [Background] Witthoft M, Rist F, Bailer J. Abnormalities in cognitive-emotional information processing in idiopathic environmental intolerance and somatoform disorders. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):70-84. doi: 10.1016/j.jbtep.2008.04.002. Epub 2008 May 23. PMID 18501333
- [Derived] Senger K, Rubel JA, Kleinstauber M, Schroder A, Kock K, Lambert MJ, Lutz W, Heider J. Symptom change trajectories in patients with persistent somatic symptoms and their association to long-term treatment outcome. Psychother Res. 2022 Jun;32(5):624-639. doi: 10.1080/10503307.2021.1993376. Epub 2021 Oct 29. PMID 34711141
- [Derived] Schwarz J, Rief W, Radkovsky A, Berking M, Kleinstauber M. Negative affect as mediator between emotion regulation and medically unexplained symptoms. J Psychosom Res. 2017 Oct;101:114-121. doi: 10.1016/j.jpsychores.2017.08.010. Epub 2017 Aug 10. PMID 28867416
- [Derived] Kleinstauber M, Gottschalk J, Berking M, Rau J, Rief W. Enriching Cognitive Behavior Therapy with Emotion Regulation Training for Patients with Multiple Medically Unexplained Symptoms (ENCERT): Design and implementation of a multicenter, randomized, active-controlled trial. Contemp Clin Trials. 2016 Mar;47:54-63. doi: 10.1016/j.cct.2015.12.003. Epub 2015 Dec 4. PMID 26655432